CLINICAL TRIAL: NCT01578304
Title: Phase IV Study to Evaluate the Efficacy and Safety Imidafenacin Versus Fesoterodine in Patients With Overactive Bladder
Brief Title: Comparison of Efficacy and Safety Between Imidafenacin and Fesoterodine in Patients With Overactive Bladder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Collaborators: Kyorin Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG-IFCL002
Record Dates: First submitted 2012-04-12; First posted 2012-04-16 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Overactive Bladder
Keywords: Overactive bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — imidafenacin; fesoterodine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imidafenacin (Experimental)
  Interventions: Drug: Imidafenacin
- Fesoterodine (Active Comparator)
  Interventions: Drug: Fesoterodine

INTERVENTIONS:
Drug: Imidafenacin — Tablet, 12 weeks twice daily
  Arms: Imidafenacin
Drug: Fesoterodine — Tablet, 12 weeks once daily
  Arms: Fesoterodine

SUMMARY:
To evaluate the efficacy and safety after 12 weeks oral administration of Imidafenacin 0.1mg b.i.d versus Fesoterodine 4mg once daily for the urge incontinence and/or increased urinary frequency associated with urgency as may occur in patients with overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with overactive bladder aged 20 years or more
* subject who had the continuos symptom for 3 months or more
* subject prepare a symptom diary and was deemed eligible for the study by the investigator
* 8 times or more of daily mean urination frequency
* 2 times or more of daily mean frequency of a sense of urinary urgency or 2 times or more of urge incontinence frequency

Exclusion Criteria:

* subjects with clinically significant stress urge incontinence, patients with urinary tract infections or relapsing urinary tract infections who had received treatment more than 4 times in the previous year
* subjects with diseases prohibiting anti-cholinergics from administration
* subjects who used an indwelling catheter or intermittent self intubation program, patients who had prostatic hyperplasia, prostatic cancer, bladder cancer,bladder stones, interstitial cystitis as complications
* subjects who received lower urinary tract surgery within 6 months
* subjects with a catheter placed or intermittent catheterization
* subjects who were deemed ineligible for the study by the investigator or sub-investigator, pregnant women, nursing women, and women who are planning pregnancy or have not used proper contraceptives during the study period
* subjects who are within 1 month after other clinical study was completed
* subjects having 100mL or more of residual urine
* subjects who had acute urinary retention history
* subjects who have been administered Prohibited concomitant medications

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2010-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Difference in daily mean urination frequency between the end of treatment period(Week 12) and the end of observation period(Baseline, Week 0) | up to 12 weeks

SECONDARY OUTCOMES:
Difference in daily mean Urinary incontinence frequency between each evaluation time(treatment period Week 4, Week 8, Week 12) and the end of observation period(Baseline, week 0) | up to 12 weeks
Difference in daily mean urge incontinence frequency between each evaluation time(treatment period Week 4, Week 8, Week 12) and the end of observation period(Baseline, week 0) | up to 12 weeks
Difference in daily mean nocturia frequency between each evaluation time(treatment period Week 4, Week 8, Week 12) and the end of observation period(Baseline, week 0) | up to 12 weeks
Difference in daily mean urination frequency between each evaluation time(treatment period Week 4, Week 8) and the end of observation period(baselien, week 0) | up to 12 weeks
Difference in QoL score between each evaluation time(treatment period Week 4, Week 8, Week 12) and the end of observation period(Baseline, week 0) | up to 12 weeks
Adverse events | up to 24 weeks
laboratory test | up to 12 weeks
vital signs | up to 12 weeks
residual urine | up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: KYU-SUNG LEE, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea